CLINICAL TRIAL: NCT01670318
Title: Study Examining the PROMUS Element Everolimus-eluting Stent in Multi-center Coronary Intervention of Complex Arterial Lesion Subsets
Acronym: SPECIALIST
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The PCI Guideline Research Society (Network)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPECIALIST Registry
Record Dates: First submitted 2012-08-16; First posted 2012-08-22 (Estimated); Last update posted 2012-08-22 (Estimated); Status verified 2012-08

CONDITIONS: Coronary Artery Disease
Keywords: Chronic total occlusion; Bifurcation lesion; Left main trunk lesion; Small vessel disease; Multi vessel disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- platinum chromium everolimus-eluting stent (Experimental)
  Interventions: Device: platinum chromium everolimus-eluting stent (PROMUS Element by Boston Scientific, Massachusetts)

INTERVENTIONS:
Device: platinum chromium everolimus-eluting stent (PROMUS Element by Boston Scientific, Massachusetts)

SUMMARY:
Randomized trials have demonstrated an excellent safety and efficacy profile for the chromium everolimus-eluting stent. The platinum chromium everolimus-eluting sten (PtCr-EES) uses the identical antiproliferative agent and polymer but with a novel platinum chromium scaffold designed for enhanced deliverability, vessel conformability, side-branch access, radiopacity, radial strength, and fracture resistance. However, the efficacy of the PtCr-EES for complex coronary artery diseases subsets such as chronic total occlusion, bifurcation lesion, left main trunk disease, and small vessel diseases is still unknown.

ELIGIBILITY:
Inclusion Criteria:

1. A patient with ischemic heart disease including stable angina pectoris and acute coronary syndrome
2. Male or non-pregnant female
3. Key lesion inclusion criteria as follows

   1. Multi-vessel diseases
   2. Long lesion (lesion length >30mm by visual estimation)
   3. Small vessel disease (reference diameter <2.5mm by visual estimation)
   4. Bifurcation lesion
   5. Ostial lesion
   6. Calcified lesion
   7. Protected or non-protected left main trunk disease
   8. Chronic total occlusion
   9. In stent restenosis of bare metal stent or everolimus-eluting stent

Exclusion Criteria:

1. Hypersensitivity to cobalt chromium, everolimus, heparin, aspirin, ticlopidine, clopidogrel or X-ray contrast media.
2. Serum creatinine level >3.0 mg/dL
3. Other concomitant disease or medical condition that could impact patient/procedural outcomes, such as history of bleeding diathesis or cancer within 5 years.

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2012-08; Primary Completion 2013-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Major adverse cardiac event including cardiac death, myocardial infarction, and target vessel revascularization | 12 month

SECONDARY OUTCOMES:
Successful stent delivery with final percent diameter stenosis less than 50% at minimum lumen diameter site | In hospital
Target lesion revascularization | 12 month
Target vessel revascularization | 12 month
Myocardial infarction | 24 month
Cardiac death | 24 month
Major adverse cardiac event including cardiac death, myocardial infarction, and target vessel revascularization | 24 month
Stent thrombosis (acute, sub-acute, late,and very late) defined by Academic Research Consortium (ARC) | 24 month

CONTACTS AND LOCATIONS:
Overall Officials: Yuji Oikawa, MD, PhD, Principal Investigator — The Cardiovascular Institute; Kenya Nasu, MD, FACC, Principal Investigator — Toyohashi Heart Center
Locations (38):
- Japan (38):
  - Aichi Medical University Hospital, Nagakute, Aichi-ken
  - Toyohashi Heart Center, Toyohashi, Aichi-ken
  - Juntendo University Urayasu Hospital, Urayasu, Chiba
  - Saiseikai Fukuoka General Hospital, Fukuoka, Fukuoka
  - Kokura Memorial Hospital, Kitakyushu, Fukuoka
  - Hoshi General Hospital, Kōriyama, Fukushima
  - Southern Tohoku Research Institute for Neuroscience, Kōriyama, Fukushima
  - Gunma Prefectural Cardiovascular Center, Maebashi, Gunma
  - Gunma University Hospital, Maebashi, Gunma
  - Ota Memorial Hospital, Ōta, Gunma
  - Megumino Hospital, Eniwa, Hokkaido
  - JA Hokkaido Engaru Kosei General Hospital, Monbetsu, Hokkaido
  - Nayoro City General Hospital, Nayoro, Hokkaido
  - Sapporo Cardio Vascular Clinic, Sapporo, Hokkaido
  - Kansai Rosai Hospital, Amagasaki, Hyōgo
  - Kakogawa East City Hospital, Kakogawa, Hyōgo
  - Kobe University Hospital, Kobe, Hyōgo
  - Tsukuba Medical Center Hospital, Tsukuba, Ibaragi
  - Yokohama Rosai Hospital, Yokohama, Kanagawa
  - Yokohama City Minato Red Cross Hospital, Yokohama, Kanagawa
  - Saiseikai Kumamoto Hospital, Kumamoto, Kumamoto
  - Daini Okamoto General Hospital, Uji, Kyoto
  - Matsumoto Kyoritsu Hospital, Matsumoto, Nagano
  - Rinku General Medical Center, Izumisano, Osaka
  - Hokusetsu General Hospital, Takatsuki, Osaka
  - SHUWA General Hospital, Kasukabe, Saitama
  - Kasukabe Chuo General Hospital, Kasukabe, Saitama
  - TODA CHUO General Hospital, Toda, Saitama
  - Seirei Mikatahara General Hospital, Hamamatsu, Shizuoka
  - Ayase Heart Hospital, Adachi-ku, Tokyo
  - Tokyo Rinkai Hospital, Edogawa-ku, Tokyo
  - Itabashi Chuo Medical Center, Itabashi-ku, Tokyo
  - Katsushika Medical Center, Katsushika-ku, Tokyo
  - Tokyo-Kita Social Insurance Hospital, Kita-ku, Tokyo
  - The Cardiovascular Institute, Minato-ku, Tokyo
  - Tokyo Metropolitan Police Hospital, Nakano-ku, Tokyo
  - Tokyo Metropolitan Hiroo Hospital, Shibuya-ku, Tokyo
  - NTT Medical Center Tokyo, Shinagawa-ku, Tokyo